CLINICAL TRIAL: NCT00943397
Title: A Multicenter, Open-Label, Controlled, Extended Safety Study of Montelukast in Infants and Young Children With Chronic Asthma
Brief Title: Extended Safety Study of Montelukast in Infants and Young Children With Chronic Asthma (0476-232)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0476-232; MK0476-232; 2009_619
Record Dates: First submitted 2009-07-21; First posted 2009-07-22 (Estimated); Results first posted 2010-06-17 (Estimated); Last update posted 2022-02-03 (Actual); Status verified 2022-02

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — montelukast

ARMS (2):
- 1 (Experimental): Montelukast
  Interventions: Drug: montelukast sodium
- 2 (Active Comparator): Usual Care
  Interventions: Drug: Comparator: Usual Care

INTERVENTIONS:
Drug: montelukast sodium — Montelukast 4 mg oral granules mixed with 1 tablespoon soft food once daily at bedtime for 52 weeks
  Other Names: Montelukast
  Arms: 1
Drug: Comparator: Usual Care — Usual care defined as inhaled/nebulized cromolyn or inhaled nedocromil or inhaled/nebulized corticosteroids, according to the investigator's usual clinical practice for 52 weeks
  Arms: 2

SUMMARY:
Patients were treated with either montelukast 4 mg oral granules or usual care. Patients who completed Protocol MK0476-176-01 (NCT00943683) had the option to enroll in this study. Additionally, patients with asthma who were 6 to 11 months of age and who had not participated in Protocol MK0476-176-01, could also enroll.

ELIGIBILITY:
Inclusion Criteria:

* Patient successfully completed visit 5 of MK0476 Protocol 176 (NCT00943683)

OR:

* Patient is in good, stable health
* Patient has been fed solid foods for at least 1 month
* Patients had at least 3 episodes of asthma or asthma-like symptoms, all occurring after 8 weeks of age; at least one within 6 months of the Prestudy Visit
* Patients had to be in need of a controller therapy according to criteria established in the Global Initiative for Asthma (GINA) guidelines

Exclusion Criteria:

* Patient was hospitalized at the start of the study or had any major surgery 4 weeks prior
* Patient had an allergy to apples or applesauce

Ages: 6 Months to 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 190 (Actual)
Dates: Start 2001-04; Primary Completion 2001-10 (Actual); Study Completion 2001-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Result] Bisgaard H, Skoner D, Boza ML, Tozzi CA, Newcomb K, Reiss TF, Knorr B, Noonan G. Safety and tolerability of montelukast in placebo-controlled pediatric studies and their open-label extensions. Pediatr Pulmonol. 2009 Jun;44(6):568-79. doi: 10.1002/ppul.21018. PMID 19449366

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited at 27 sites in Africa, Europe, North America, and South America Therapy period: May 2001 to Mar 2003.
Pre-assignment Details: This was an open-label, controlled extended safety study. Patients were treated with either montelukast 4-mg oral granules or usual care. Patients who completed Protocol 176-01 had the option to enroll in this study. Additionally, patients with asthma who were 6 to 11 months of age and who had not participated in Protocol 176-01, could also enroll.
Groups:
- Usual Care: Usual care: defined as inhaled/nebulized cromolyn or inhaled nedocromil or inhaled/nebulized corticosteroids, according to the investigator's usual clinical practice for 52 weeks
- Montelukast: Montelukast 4-mg oral granules mixed with 1 tablespoon soft food once daily at bedtime for 52 weeks.
Period: Overall Study
Arm/Group | Usual Care | Montelukast
Started | 32 | 158
Completed | 17 (Site terminated - Merck administrative decision (11); Discontinued for other (1)) | 86 (Site terminated - Merck administrative decision (52); Patient moved (1); Discontinued for other (3))
Not Completed | 15 | 72
Not completed — Adverse Event | 0 | 6
Not completed — Lost to Follow-up | 0 | 4
Not completed — Protocol Violation | 2 | 5
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Site terminated and other | 12 | 56

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Usual Care | Montelukast | Total
Number analyzed (Participants) | 32 | 158 | 190
Age, Continuous [Mean (Standard Deviation); unit: Months] | 16.69 (7.22) | 16.45 (7.41) | 16.49 (7.36)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 45 | 56
  Male | 21 | 113 | 134

OUTCOME MEASURES:

1. Primary Outcome: Number of Clinical Adverse Experiences (CAEs) Reported by Patients With up to 52 Weeks of Treatment
Description: An adverse experience (AE) is defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally associated with the use of the SPONSOR'S product, whether or not considered related to the use of the product
Time Frame: Up to 52 weeks of treatment
Population: All patients who took study medication were included in the analysis.
Measure: Number; unit: Participants
Arm/Group | Usual Care | Montelukast
Number analyzed (Participants) | 32 | 158
Participants
  With CAEs | 31 | 156
  Without CAEs | 1 | 2

ADVERSE EVENTS:
Time Frame: Over 52 weeks of treatment and including 14 days follow-up post-treatment AE
Arm/Group | Usual Care | Montelukast
Serious Adverse Events (participants affected / at risk) | 1/32 | 15/158
Other Adverse Events (participants affected / at risk) | 30/32 | 155/158
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Usual Care (N=32) | Montelukast (N=158)
Bacterial Infection (Infections and infestations) | 0 | 3
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Diarrhea (Gastrointestinal disorders) | 1 | 0
Enteritis (Gastrointestinal disorders) | 0 | 1
Gastroenteritis (Gastrointestinal disorders) | 0 | 1
Parotitis (Gastrointestinal disorders) | 0 | 1
Laryngitis (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pharyngitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Tonsillar Disorder (General disorders) | 0 | 2
Tonsillitis (Infections and infestations) | 0 | 1
Seizure (Nervous system disorders) | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Laryngotracheitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Usual Care (N=32) | Montelukast (N=158)
Bacterial Infection (Infections and infestations) | 2 | 4
Fever (General disorders) | 7 | 26
Influenza-Like Disease (General disorders) | 2 | 20
Upper Respiratory Infection (Infections and infestations) | 15 | 82
Viral Infection (Infections and infestations) | 9 | 17
Diarrhea (Gastrointestinal disorders) | 8 | 30
Gastroenteritis (Gastrointestinal disorders) | 2 | 9
Vomiting (Gastrointestinal disorders) | 3 | 10
Allergic Rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 | 19
Conjunctivitis (Eye disorders) | 3 | 15
Nasopharyngeal Disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 12
Otitis (Ear and labyrinth disorders) | 3 | 1
Otitis Media (Ear and labyrinth disorders) | 7 | 39
Pharyngitis (Respiratory, thoracic and mediastinal disorders) | 14 | 58
Rhinitis (Respiratory, thoracic and mediastinal disorders) | 3 | 18
Sinusitis (Respiratory, thoracic and mediastinal disorders) | 2 | 11
Tonsillitis (Infections and infestations) | 1 | 9
Asthma (Respiratory, thoracic and mediastinal disorders) | 18 | 77
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 7 | 22
Pneumonia (Infections and infestations) | 1 | 9
Respiratory Infection (Infections and infestations) | 1 | 9
Contact Dermatitis (Skin and subcutaneous tissue disorders) | 2 | 1
Cutaneous Candidiasis (Infections and infestations) | 3 | 6
Eczematous Dermatitis (Skin and subcutaneous tissue disorders) | 4 | 12
Varicella (Infections and infestations) | 3 | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Merck agreements may vary with individual investigators, but will not prohibit any investigator from publishing. Merck supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.